CLINICAL TRIAL: NCT03125889
Title: Acute Hemostasis Following the Use of the AQUABEAM® System for the Treatment of Benign Prostatic Hyperplasia II
Acronym: AHA II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP0131
Record Dates: First submitted 2017-03-14; First posted 2017-04-24 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Image-guided; BPH; Aquablation; AQUABEAM; LUTS; Tissue resection; Robotics
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Arm (Experimental): Subjects will receive treatment with the AquaBeam System to remove prostatic tissue.
  Interventions: Device: AquaBeam System

INTERVENTIONS:
Device: AquaBeam System — The AquaBeam system delivers a high-velocity saline stream under precise electromechanical control and live ultrasound guidance to ablate prostatic glandular tissue without the production of heat. The physician uses ultrasound imaging to plan the treatment contour and depth to define the treatment region. The AquaBeam ablates the target tissue, adhering to the pre-defined treatment zone.

SUMMARY:
A single-arm prospective, interventional clinical trial to evaluate the safety and performance of obtaining hemostasis following prostate resection using the AQUABEAM for treatment of LUTS resulting from BPH.

DETAILED DESCRIPTION:
PROCEPT BioRobotics has developed the AQUABEAM, a personalized image-guided waterjet resection system that utilizes a high-velocity saline stream to resect and remove prostate tissue in males suffering from LUTS due to BPH. The AQUABEAM System is intended for the resection and removal of prostate tissue in patients experiencing lower urinary tract symptoms (LUTS).The primary objective of this study is to evaluate the safety and performance of obtaining hemostasis with catheters following prostate resection using AQUABEAM for the treatment of LUTS resulting from BPH. Up to 50 participants will be included in the trial at one clinical study site. All patients will be followed up for 30 days for safety assessment prior to study exit. The trial is a single-arm prospective, interventional clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male
* BPH symptoms

Exclusion Criteria:

* Serious concurrent medical conditions

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Completion of the intended surgical procedure with adequate hemostasis | 7 days post-op
Proportion of subjects who return to the OR for bleeding treatment or requires transfusion | 7 days post-op

CONTACTS AND LOCATIONS:
Locations (1):
- Muljibhai Patel Urological Hospital, Nadiād, Gujarat, India

IPD SHARING:
Plan to Share IPD: Undecided